CLINICAL TRIAL: NCT06111144
Title: Effects of Polarized and Pyramidal Training Models Combined With or Without Mindfulness on Running Time, Performance Variables, and Body Composition in Amateur Long-distance Runners. A Randomized Controlled Trial
Brief Title: Effects of Polarized and Pyramidal Training Combined With or Without Mindfulness in Amateur Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victor Hugo Arboleda Serna, Principal Investigator, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TID-Runners-UdeA-JCRunning
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Training intensity distribution; Polarized training; Pyramidal training; Amateur long-distance runners

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Polarized training Intensity distribution model without mindfulness program (Experimental): The TID of the entire training program will be zone 1 (80%), zone 2 (5%), zone 3 (15%).
  The periodization of the training will be performed in a 3:1 load-recovery cycle, that is, three weeks of load for one week of recovery, this cycle will be repeated 3 times to complete the 12 weeks. The running sessions will have a volume in the load weeks as follows: The first week a volume of 5 hours, the second week 5.5 hours and the third week 6 hours. In the recovery week the volume will be 4 hours. As for the running technique and strength, these will have a weekly volume of 30 min and 1 hour respectively during all 12 weeks.
  In summary:
  60 running sessions 24 strength sessions 24 running technique sessions
  Interventions: Behavioral: Polarized training intensity distribution (TID) without mindfulness
- Pyramidal training Intensity distribution model without mindfulness program (Experimental): The TID of the entire training program will be zone 1 (80%), zone 2 (5%), zone 3 (15%).
  The periodization of the training will be performed in a 3:1 load-recovery cycle, that is, three weeks of load for one week of recovery, this cycle will be repeated 3 times to complete the 12 weeks. The running sessions will have a volume in the load weeks as follows: The first week a volume of 5 hours, the second week 5.5 hours and the third week 6 hours. In the recovery week the volume will be 4 hours. As for the running technique and strength, these will have a weekly volume of 30 min and 1 hour respectively during all 12 weeks.
  In summary:
  60 running sessions 24 strength sessions 24 running technique sessions
  Interventions: Behavioral: Pyramidal training intensity distribution (TID) without mindfulness
- Polarized training Intensity distribution model with mindfulness program (Experimental): The TID of the entire training program will be zone 1 (80%), zone 2 (5%), zone 3 (15%).
  The periodization of the training will be performed in a 3:1 load-recovery cycle, that is, three weeks of load for one week of recovery, this cycle will be repeated 3 times to complete the 12 weeks. The running sessions will have a volume in the load weeks as follows: The first week a volume of 5 hours, the second week 5.5 hours and the third week 6 hours. In the recovery week the volume will be 4 hours. As for the running technique, strength and mindfulness these will have a weekly volume of 30 min, 1 hour and 65 min respectively during all 12 weeks.
  The weekly mindfulness practice will be done in 4 different types of sessions: (life-meditation, jogging-meditation, stretching-meditation, running-meditation).
  In summary:
  60 running sessions 60 mindfulness sessions 24 strength sessions 24 running technique sessions
  Interventions: Behavioral: Polarized training intensity distribution (TID) and mental training using mindfulness
- Pyramidal training Intensity distribution model with mindfulness program (Experimental): The TID of the entire training program will be zone 1 (80%), zone 2 (15%), zone 3 (5%).
  The periodization of the training will be performed in a 3:1 load-recovery cycle, that is, three weeks of load for one week of recovery, this cycle will be repeated 3 times to complete the 12 weeks. The running sessions will have a volume in the load weeks as follows: The first week a volume of 5 hours, the second week 5.5 hours and the third week 6 hours. In the recovery week the volume will be 4 hours. As for the running technique, strength and mindfulness these will have a weekly volume of 30 min, 1 hour and 65 min respectively during all 12 weeks.
  The weekly mindfulness practice will be done in 4 different types of sessions: (life-meditation, jogging-meditation, stretching-meditation, running-meditation).
  In summary:
  60 running sessions 60 mindfulness sessions 24 strength sessions 24 running technique sessions
  Interventions: Behavioral: Pyramidal training intensity distribution (TID) and mental training using mindfulness

INTERVENTIONS:
Behavioral: Polarized training intensity distribution (TID) and mental training using mindfulness — Polarized TID model group with mindfulness program (POL+)
  Arms: Polarized training Intensity distribution model with mindfulness program
Behavioral: Pyramidal training intensity distribution (TID) and mental training using mindfulness — Pyramidal TID model group with mindfulness program (PYR+)
  Arms: Pyramidal training Intensity distribution model with mindfulness program
Behavioral: Polarized training intensity distribution (TID) without mindfulness — Polarized TID model group without mindfulness program (POL-)
  Arms: Polarized training Intensity distribution model without mindfulness program
Behavioral: Pyramidal training intensity distribution (TID) without mindfulness — Pyramidal TID model group without mindfulness program (PYR-).
  Arms: Pyramidal training Intensity distribution model without mindfulness program

SUMMARY:
Road running in athletics has grown worldwide in recent years, which has led to an increase in the number of recreational runners. Despite this growth, research addressing this population is scarce, with major limitations and methodological weaknesses. Two of the topics of recent interest in runners are the effects of training intensity distribution (TID) and mental training using mindfulness on running time, body composition and physiological parameters related to performance in endurance sports; the maximal oxygen consumption (VO2max), maximal aerobic speed (MAS) and ventilatory thresholds (VT).

The scarce evidence found identifies the TID polarized model as the most effective in sports performance and TID pyramidal model as the most used by elite runners. For mindfulness, it is identified as an emerging program that could contribute to performance in endurance sports.

DETAILED DESCRIPTION:
40 recreational long-distance runners will be randomly assigned into one of the following 4 TID models groups: polarized TID model group with mindfulness program (POL+), polarized TID model group without mindfulness program (POL-), pyramidal TID model group with mindfulness program (PYR+) and pyramidal TID model group without mindfulness program (PYR-). Each group will be composed of 10 subjects. The interventions will have a duration of 12 weeks.

All participants will have evaluation of 10 km running time, body composition and physiological parameters (VO2max, MAS and VT's 1 and 2) at week 0 and 13 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Amateur long-distance runners
* Running time of 10 km in Bogotá, Colombia or similar altitude (2600 m above sea level) for men between 45 and 60 minutes, and for women between 50 and 65 minutes.

Exclusion Criteria:

* Smokers.
* History of cardiovascular disease.
* Arrhythmias.
* Cardiac insufficiencies.
* Hypertension.
* Musculoskeletal problems that affect their participation in the training program.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in 10 km race time | Week 0 and 13
  The time in the 10 km will be taken by two evaluators with independent stopwatches, and the average of them will be taken as the official time. The test will take place in a 1257 m loop, with a positive difference in altitude of 5 m.

SECONDARY OUTCOMES:
Change in VO2max | Week 0 and 13
  Incremental test to exhaustion on a Woodway© model 4Front treadmill. During the test, VO2 will be measured breath-by-breath by a portable metabolic system COSMED© model K5.
  The VO2max will be calculated as the average oxygen consumption of the last 30 seconds measured in the incremental test.
Change in ventilatory threshold 1 | Week 0 and 13
  Incremental test to exhaustion on a Woodway© model 4Front treadmill. During the test, ventilatory threshold 1 will be measured by a portable metabolic system COSMED© model K5.
  Ventilatory threshold 1 will be defined as the first increase in ventilatory equivalent for oxygen (VE/VO2) vs. load, without a simultaneous increase in ventilatory equivalent for carbon dioxide (VE/VCO2) vs. load.
Change in ventilatory threshold 2 | Week 0 and 13
  Incremental test to exhaustion on a Woodway© model 4Front treadmill. During the test, ventilatory threshold 2 will be measured by a portable metabolic system COSMED© model K5.
  Ventilatory threshold 2 will be defined as the second increase in ventilation with a concomitant rapid increase in VE/VO2 and VE/VCO2 and a decrease in the partial pressure of exhaled carbon dioxide (PETCO2).
Change in maximal aerobic speed | Week 0 and 13
  Incremental test to exhaustion on a Woodway© model 4Front treadmill. During the test, maximal aerobic speed will be measured by a portable metabolic system COSMED© model K5.
  The maximal aerobic speed will be determined at the speed corresponding to the VO2max.
Change in body weight | Week 0 and 13
  Body weight (kg) will be obtained using a HBF-514C OMRON© body composition analyzer
Change in body fat | Week 0 and 13
  Body fat (%) will be obtained using a HBF-514C OMRON© body composition analyzer
Change in muscle mass | Week 0 and 13
  Muscle mass (%) will be obtained using a HBF-514C OMRON© body composition analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- JC Running, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No